CLINICAL TRIAL: NCT06844929
Title: Suleyman Demirel University Health Sciences Faculty
Brief Title: Impact of Podcast-Based Breastfeeding Education During Pregnancy on Breastfeeding Self-Efficacy in Pregnant Women
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Suleyman Demirel University (Other)
Responsible Party: Principal Investigator, İlknur Atasever, Assistant Professor, Suleyman Demirel University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: BREASTFEED_PODCAST_2024; Suleyman Demirel University (Other: Suleyman Demirel University)
Record Dates: First submitted 2025-02-12; First posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Pregnant Women; Breastfeeding
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: statistician
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Podcast Group (Experimental): Creating the content of podcast-based training Obtaining expert opinions on the content Recording podcasts at the Radio Television Application and Research Center
  Interventions: Other: Podcast Group
- Brochure Group (Other): Preparation of brochures for breastfeeding education Obtaining expert opinions
  Interventions: Other: Brochure Group

INTERVENTIONS:
Other: Podcast Group — Providing breastfeeding education via podcast
  Arms: Podcast Group
Other: Brochure Group — Providing standard breastfeeding education using brochures
  Arms: Brochure Group

SUMMARY:
Women who meet the sampling selection criteria will be introduced and informed about the study. Considering the patients who meet the research criteria and accept the study, patients will be divided into groups according to whether their barcode numbers are odd or even (1:1 ratio), provided that the number of individuals in the intervention and control groups is equal. It is planned to work with a total of 80 pregnant women, considering the losses. The intervention and control groups will be selected by drawing lots. The Introductory Information Form and Prenatal Breastfeeding Self-Efficacy Scale will be filled out by the women who meet the sampling selection criteria and accept to participate in the study before the application. The content of the podcast-based education to be given to the pregnant women in the intervention group will be created by the researcher and the consultant, and expert opinion will be obtained regarding the content. For the pregnant women in the control group; a brochure will be prepared for breastfeeding education and expert opinion will be obtained. The brochure prepared by the researcher and the consultant will be given to the pregnant women in the control group at the planned time. The pregnant women in the intervention group will be given a period of two weeks to complete the prepared podcast education. At the end of the two-week period, pregnant women in the intervention and control groups will be asked to fill out the Prenatal Breastfeeding Self-Efficacy Scale again.

DETAILED DESCRIPTION:
Location of the study: The study is planned to be conducted in the Obstetrics Department of Süleyman Demirel University, Faculty of Medicine. The Department of Gynecology and Obstetrics was established in 1994 in the old faculty of medicine hospital in the city center. Over time, with its 5 outpatient clinic rooms and 38-bed capacity, it has become an important reference center in the Lakes Region and its surroundings, especially in complicated patient approaches. Süleyman Demirel University, Faculty of Medicine, Department of Gynecology and Obstetrics contributes to health services with its faculty members specialized in General Gynecology, Obstetrics, High Risk Pregnancies, Infertility, Assisted Reproductive Techniques (IVF), Gynecologic Oncology, Gynecologic Endoscopic Surgery, Urogynecology. Time of the study: The study will be conducted between April 2024 and January 2025. Research universe, sample, research group: The research universe will consist of women who voluntarily accept to participate in the study and apply to the Obstetrics and Gynecology outpatient clinic of Süleyman Demirel University Research and Practice Hospital. The criteria for inclusion in the study are as follows: • Being literate and speaking Turkish • Agreeing to participate in the research Research method and data collection tools: The data of this study will be collected with the Descriptive Characteristics Form and the Prenatal Breastfeeding Self-Efficacy Scale. Descriptive Characteristics Form: It will be developed by the researchers and will include questions about some sociodemographic data of the pregnant women and their breastfeeding experiences. The Prenatal Breastfeeding Self-Efficacy Scale was developed by Wells et al. in 2006 in order to determine the breastfeeding self-efficacy perceptions of pregnant women in the prenatal period. The scale consists of a total of 20 items (Appendix-III). The original scale has a total of 4 sub-dimensions. These are: Skills and Desires Sub-dimension: It consists of a total of 7 items. These items are items 6, 7, 8, 9, 10, 11 and 12. The lowest score that can be obtained from this subdimension is 7 and the highest score is 35. Information Acquisition Subdimension: It consists of a total of 5 items. These items are items 1, 2, 3, 5 and 17. The lowest score that can be obtained from this subdimension is 5 and the highest score is 25. Viewpoint of Surrounding People Subdimension: It consists of a total of 4 items. These items are items 13, 14, 15 and 16. The lowest score that can be obtained from this subdimension is 4 and the highest score is 20. Social Pressure Subdimension: It consists of a total of 2 items. These items are items 18 and 19. The lowest score that can be obtained from this subdimension is 2 and the highest score is 10. The validity and reliability of the scale for Turkish was made by Aydın and Pasinlioğlu in 2016 (Aydın & Pasinlioğlu., 2018). Implementation of the Study: Women who meet the sampling selection criteria will be met and informed about the study. Considering the patients who meet the research criteria and accept the study, the patients will be divided into groups according to whether their barcode numbers are odd or even, provided that the number of individuals in the intervention and control groups is equal (1:1 ratio). It is planned to work with a total of 80 pregnant women, considering the losses. The intervention and control groups will be selected by drawing lots. The Introductory Information Form and Prenatal Breastfeeding Self-Efficacy Scale will be filled out by the women who meet the sampling selection criteria and accept to participate in the study before the application. The content of the podcast-based education to be given to the pregnant women in the intervention group will be created by the researcher and the consultant, and expert opinion will be obtained regarding the content. For the pregnant women in the control group; a brochure will be prepared for breastfeeding education and expert opinion will be obtained. The brochure prepared by the researcher and the consultant will be given to the pregnant women in the control group at the planned time. The pregnant women in the intervention group will be given a period of two weeks to complete the prepared podcast education. At the end of the two-week period, pregnant women in the intervention and control groups will be asked to fill out the Prenatal Breastfeeding Self-Efficacy Scale again.

Education Content: Benefits of breastfeeding, How breastfeeding mothers should be fed Hormones, What to consider when breastfeeding, Breastfeeding problems, Symptoms of insufficient milk, Reasons for and treatment of breast refusal,Necessary information on storing breast milk. Evaluation of Data: Data evaluation will be done in a computer environment using SPSS (Statistical Package For Social Sciences) 21.0 package program. Percentage distributions, mean, standard deviation chi-square test, t-test in dependent groups will be used in the analysis of data. Research findings will be evaluated at a 95% confidence interval and at a significance level of p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Be primiparous
* To consent to participate in the research.

Exclusion Criteria:

-Not completing any stage of the study

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-09-15 (Actual); Primary Completion 2025-03-21 (Estimated); Study Completion 2025-03-21 (Estimated)

PRIMARY OUTCOMES:
Measuring the effect of podcast-based breastfeeding education on pregnant women's Prenatal Breastfeeding Self-Efficacy Scale scores. | Before the intervention and 2 weeks after completing the podcast training
  The differences in Prenatal Breastfeeding Self-Efficacy Scale scores between women who received podcast-based breastfeeding education and those who received brochure-based breastfeeding education will be evaluated.The total score on the Prenatal Breastfeeding Self-Efficacy Scale ranges from a minimum of 20 to a maximum of 100. Higher scores indicate greater breastfeeding self-efficacy

CONTACTS AND LOCATIONS:
Overall Officials: İlknur Atasever, Dr., Principal Investigator — Suleyman Demirel University
Locations (1):
- İlknur Atasever, Isparta, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Our plan aims to ensure transparent sharing of research results and accessibility to the scientific community. Individual participant data will be safeguarded in accordance with privacy standards